CLINICAL TRIAL: NCT03726606
Title: A Randomized, Controlled, Two-armed, and Single Blind Trial Evaluating the Visual Performance and Quality of Vision After Bilateral Implantation of 2 Presbyopia Correcting Intraocular Lenses: Trifocal Versus Extended Depth of Focus
Brief Title: A Comparison of the Visual Performance of Trifocal Versus Extended Depth of Focus Intraocular Lenses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hashmanis Hospital (Other)
Collaborators: SIFI SpA (Industry); Hashmanis Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HASH00011
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Cataract; Lenses; Visual Impairment
Keywords: Cataract; Intraocular lenses; Trifocal intraocular lenses; Extended depth of focus intraocular lenses; Presbyopia
MeSH Terms: conditions — Cataract; Vision Disorders; Presbyopia | interventions — Lenses, Intraocular

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of two arms: Trifocal or extended depth of focus intraocular lenses.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the examiner will be blinded to the arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended depth of focus intraocular lens (Experimental): Bilateral implantation of extended depth of focus intraocular lenses.
  Interventions: Device: Intraocular lens
- Trifocal intraocular lens (Active Comparator): Bilateral implantation of trifocal intraocular lenses.
  Interventions: Device: Intraocular lens

INTERVENTIONS:
Device: Intraocular lens — Bilateral implantation of the same intraocular lens.
  Other Names: Phacoemulsifcation

SUMMARY:
We are conducting a trial evaluating the performance of trifocal versus extended depth of focus intraocular lenses. These lenses will be implanted in otherwise healthy individuals with visual problems due to bilateral cataracts. Patients must be seeking an improvement in their visual performance with a special focus on presbyopia correction.

DETAILED DESCRIPTION:
To compare the clinical performance, quality of vision and subjective outcomes between the extended depth of focus (EDOF) Mini Well Ready intraocular lens (IOL) and the diffractive trifocal PanOptix IOL, at 3 months following second eye implantation.

Statistical analysis

All data will be analyzed using the Statistical Package for the Social Sciences (SPSS) v23 (SPSS Inc., Chicago, IL, USA). Graphs will be made using SPSS and Microsoft Excel (Microsoft Corp., Redmond, WA, USA). Normality will be tested for using the Shapiro Wilk test. If the data is normal, an independent t test will be used for comparing the continuous variables between the groups. If the data is not normal, then we will utilize the Mann Whitney U test.

Sample size calculation

The sample size calculation was based on the mean binocular Uncorrected Near Visual Acuity (UNVA) tested at 40cm under photopic condition. A previous study on the same diffractive trifocal IOL revealed a binocular UNVA of 0.01 ± 0.087 logMAR (12). The anticipated mean value for Mini Well Toric Ready is 0.10 logMAR. Based on these assumptions, an alpha of 0.05 and power of 0.8, it was calculated a number of 15 patients implanted bilaterally for each group. Assuming a dropout rate of 20% on the primary outcome measure, this resulted in a total number of 36 bilateral patients, 18 each group.

Duration of the project: Six months to one year

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 30 years of age or older
* Has bilateral cataracts with visual problems
* Is motivated for vision correction

Exclusion Criteria:

* Any ocular pathology that could impair vision, for example:

  * Pseudoexfoliation syndrome
  * Zonular weakness
  * Retinal or corneal dystrophies
  * Retinal pathologies like age related macular degeneration
* History of trauma
* History of ocular surgery
* Individuals having trouble understanding written or spoken language
* Those with dense cataracts causing problems with optical biometry
* Average corneal powers outside the range of 41 diopters (D) to 46 D
* Corneal astigmatism > 0.75 D
* Irregular astigmatism index of 0.54 or higher

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-11-05 (Estimated); Primary Completion 2019-05-06 (Estimated); Study Completion 2019-05-06 (Estimated)

PRIMARY OUTCOMES:
Near Visual Acuity (Corrected and Uncorrected) | 3 months after bilateral implantation
  40 cm
Intermediate Visual Acuity (Corrected and Uncorrected) | 3 months after bilateral implantation
  66 cm
Distance Visual Acuity (Corrected and Uncorrected) | 3 months after bilateral implantation
  4 m

SECONDARY OUTCOMES:
Defocus Curve | 3 months after bilateral implantation
  Evaluating presbyopia correction
Objective Automated Refraction | 3 months after bilateral implantation
  Using a auto refractometer (Topcon KR-800, Tokyo, Japan)
Contrast Sensitivity | 3 months after bilateral implantation
  At 2.5 m
Higher Order Abberations | 3 months after bilateral implantation
  Using a Abberometer
Halos and Glares | 3 months after bilateral implantation
  Using custom software provided by SIFI

CONTACTS AND LOCATIONS:
Overall Officials: Sharif Hashmani, FCPS, Principal Investigator — Hashmanis Hospital

IPD SHARING:
Plan to Share IPD: Undecided